CLINICAL TRIAL: NCT01939938
Title: Pilot Study of the Comparison of the Upper Airway Dynamics of Oronasal vs Nasal Masks With Positive Airway Pressure Treatment
Brief Title: Pilot Study of the Comparison of the Upper Airway Dynamics of Oronasal vs Nasal Masks With PAP Treatment
Acronym: Mask_MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1207012713
Record Dates: First submitted 2013-08-13; First posted 2013-09-11 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects-Nasal and Oronasal PAP Mask (Experimental): Each subject will be imaged in a dynamic MRI with both a oronasal and nasal mask at pressures of 5, 10, and 15 cm of H2O.
  Interventions: Device: Nasal and Oronasal PAP Mask

INTERVENTIONS:
Device: Nasal and Oronasal PAP Mask — Subjects will be imaged via MRI wearing a nasal and oronasal PAP mask at 5, 10 and 15 cm H20.

SUMMARY:
Our group has recently found that the choice of positive airway pressure mask can significantly affect the pressure required to adequately treat sleep disordered breathing. The goal of this study is to visualize the upper airway in the retropalatal and retroglossal region while using both oronasal and nasal masks with CPAP in order to investigate differences in upper airway dynamics that may occur between these two mask types.

DETAILED DESCRIPTION:
It is known that oronasal masks are not as effective at opening the upper airway compared to nasal only continuous positive airway pressure (CPAP) masks in patients with sleep-disordered breathing. However, the physiological mechanism for this difference in efficacy is not known; although, it has been hypothesized to involve the retroglossal and/or retropalatal region of the upper airway. The objective of this study was to investigate differences in retroglossal and retropalatal anterior-posterior space with the use of oronasal vs. nasal CPAP masks using real-time cine magnetic resonance imaging (cMRI).

ELIGIBILITY:
Inclusion Criteria:

* AHI> 30/hr
* 18-75 years of age

Exclusion Criteria:

* History of claustrophobia
* History of pacemaker, nerve stimulator, or any other metal implanted device

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ebben, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Center for Sleep Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ebben MR, Milrad S, Dyke JP, Phillips CD, Krieger AC. Comparison of the upper airway dynamics of oronasal and nasal masks with positive airway pressure treatment using cine magnetic resonance imaging. Sleep Breath. 2016 Mar;20(1):79-85. doi: 10.1007/s11325-015-1187-x. Epub 2015 Apr 30. PMID 25924934

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects-Nasal and Oronasal PAP Mask
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects-Nasal and Oronasal PAP Mask
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: AHI
Description: The AHI is the number of apneas or hypopneas recorded during the study per hour of sleep. It is generally expressed as the number of events per hour.
Time Frame: through study completion, an average of 1 hour
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- Baseline AHI: AHI at baseline.
- Residual AHI: AHI residual.
Arm/Group | Baseline AHI | Residual AHI
Number analyzed (Participants) | 10 | 10
events per hour | 42.3 (28.7) | 1.58 (1.87)

2. Secondary Outcome: MRI of Upper Airway With Opposite PAP Mask
Description: MRI will be used to obtain airway measurements and the position of soft tissue elements of the oropharyngeal airway will be evaluated while positive airway pressure in introduced through the opposite mask type.
Time Frame: Approximately 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects-Nasal and Oronasal PAP Mask
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Arm/Group | All Subjects-Nasal and Oronasal PAP Mask
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes